CLINICAL TRIAL: NCT06909799
Title: A Confirmatory Trial of Adjunctive N-acetylcysteine to Prevent Post Tuberculosis Lung Disease (NAC-PTLD) - A TB SEQUEL II Substudy
Brief Title: A Confirmatory Trial of Adjunctive NAC to Prevent Post Tuberculosis Lung Disease
Acronym: NAC-PTLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Research Center Borstel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AUR1-1-420
Record Dates: First submitted 2024-11-08; First posted 2025-04-04 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis (TB)
Keywords: NAC; N-acetylcysteine; HDT; Host directed therapy; PTLD; Post TB lung disease
MeSH Terms: conditions — Tuberculosis | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: NAC dosing will be 1800mg PO BID during months 1-6, or control, depending on study arm. All participants will also receive standard TB treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-Acetylcysteine (NAC) 1800mg orally twice a day plus TB treatment during months 1-6. (Experimental): N-Acetylcysteine (NAC) dosing will be 1800mg orally twice a day during months 1-6 plus standard TB treatment. This will be followed by 6 months follow up.
  Interventions: Drug: N-Acetyl Cysteine (NAC); Drug: Standard TB treatment
- Standard TB treatment during months 1-6 (Active Comparator): Standard TB treatment for 6 months followed by 6 months of observation. TB treatment will be provided as fixed dose combination tablets.
  Interventions: Drug: Standard TB treatment

INTERVENTIONS:
Drug: N-Acetyl Cysteine (NAC) — NAC will be provided as 600 mg capsules from NOW Healthgroup. Standard TB treatment will be provided as fixed dose combination tablets.
  Arms: N-Acetylcysteine (NAC) 1800mg orally twice a day plus TB treatment during months 1-6.
Drug: Standard TB treatment — Standard TB treatment will be provided as fixed dose combination tablets.

SUMMARY:
The goal of this clinical trial is to evaluate if N-acetylcysteine (NAC) works to prevent post-tuberculosis lung disease (PTLD) in patients with severe pulmonary impairment. It also aims to assess the safety of NAC. The main questions the study aims to answer are: Does NAC improve lung function (FEV1%) over 12 months in participants with pulmonary tuberculosis and baseline risk factors for PTLD? What medical issues or adverse events do participants experience while taking NAC? Researchers will compare NAC treatment to a control group to see if it can prevent PTLD when given in addition to standard TB treatment.

Participants will: Take NAC (1800mg twice daily) for 6 months with standard TB treatment or receive standard TB treatment alone; Attend scheduled clinic visits for 12 months, during which they will have respiratory assessments, blood tests, and symptom monitoring; Complete quality-of-life questionnaires and provide sputum and blood samples for analysis at multiple time points.

DETAILED DESCRIPTION:
Study Summary: This prospective, randomized, controlled, parallel-arm, open-label clinical trial evaluates the efficacy of N-acetylcysteine (NAC) as an adjunctive therapy for persons with pulmonary tuberculosis and risk factors for PTLD. The study aims to determine the long-term impact of NAC on lung function, respiratory symptoms, and quality of life in patients with drug-sensitive, culture-confirmed pulmonary tuberculosis (TB).

Study Rationale: Pulmonary TB is a leading cause of chronic lung impairment globally. PTLD results in significant morbidity even after successful TB treatment. Prior research suggests NAC may mitigate oxidative stress and preserve lung function in TB patients. This trial seeks to confirm and expand findings from the NAC-TB sub-study of TB Sequel regarding PTLD prevention and treatment.

This trial aims to provide robust evidence on the role of NAC in PTLD management, potentially informing future TB treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Persons aged 18 to 65 years
2. Willing and able to provide signed written consent, or witnessed oral con-sent with thumbprint in the case of illiteracy, prior to undertaking any trial-related procedures.
3. Body weight (in light clothing without shoes) between 30 and 90 kg.
4. Xpert TB/RIF OR Ultra showing RIF-S-MTB, with subsequent confirmation of MTB by culture.
5. Chest radiograph meeting criteria for moderate or far advanced pulmonary tuberculosis 1
6. FEV1 ≤65% of predicted adjusted for age, height, sex, and race
7. If female, of child-bearing potential and sexually active, willing to use a contraceptive method for the duration of study participation
8. HIV-1/2 seronegative, or if seropositive: CD4 T cell count ≥100/mcL and either currently receiving ART or willing to start ART during study participation

Exclusion Criteria:

1. Any condition for which participation in the trial, as judged by the investigator, could compromise the well-being of the subject or prevent, limit or confound protocol specified assessments, such as pneumothorax or clinically significant pleural effusion
2. Pregnancy or breast-feeding
3. Is critically ill, and in the judgment of the investigator has a diagnosis likely to result in death during the trial or the follow-up period.
4. TB meningitis or other forms of severe tuberculosis with high risk of a poor outcome as judged by the investigator.
5. History of allergy or hypersensitivity to any of the trial therapies or related substances, including known allergy or suspected hypersensitivity to rifampin.
6. Having participated in other clinical trials with investigational agents within 8 weeks prior to trial start or currently enrolled in an investigational trial.
7. No more than 5 days treatment for the current TB episode, and no other TB treatment in the preceding 6 months
8. Angina pectoris requiring treatment with nitroglycerin or other nitrates
9. Cardiac arrhythmia requiring medication, or any clinically significant ECG abnormality, in the opinion of the investigator
10. Random blood glucose >140 mg/dL (or >7.8 mmol/L), or history of unstable Diabetes Mellitus which required hospitalization for hyper- or hypoglycaemia within the past year prior to start of screening.
11. Use of systemic corticosteroids within the past 28 days, or a likely to require corticosteroids for management of another medical condition during the period of study participation.
12. Patients requiring treatment with medications not compatible with rifampin, such as HIV protease inhibitors
13. Subjects with any of the following abnormal laboratory values:

    1. creatinine >2 mg/dL
    2. haemoglobin <8 g/dL
    3. platelets <100x109 cells/L
    4. serum potassium <3.5
    5. aspartate aminotransferase (AST) ≥2.0 x ULN
    6. alkaline phosphatase (AP) >5.0 x ULN
    7. total bilirubin >1.5 mg/dL
    8. positive HBsAg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
FEV1% of predicted at month 12 | month 12
  Measured by spirometry

SECONDARY OUTCOMES:
FEV1% | Through study completion, an average of 12 months
  FEV1%, at other time points and as summary measures over time
FVC% | Through study completion, an average of 12 months
  FVC%, at other time points and as summary measures over time using mixed effects modeling;
FEV/FVC | Through study completion, an average of 12 months
  FEV/FVC at other time points and as summary measures over time using mixed effects modeling;
Exacerbations | Through study completion, an average of 12 months
  Number and severity of exacerbations
Respiratory QoL at multiple time points | Through study completion, an average of 12 months
  Measured using questionnaires
Respiratory symptoms | Through study completion, an average of 12 months
  Respiratory symptoms at multiple time points
Whole blood total glutathione | Through study completion, an average of 12 months
  Whole blood total glutathione at multiple time points
Mtb sputum culture | Month 2, 3 and 6
  Microbiological test that detects viable Mycobacterium tuberculosis in sputum samples
Change in MGIT (Mycobacterial Growth Indicator Tube) time to positivity (TTP): assessed over time through repeated measurements | Through study completion, an average of 12 months
  To reflect treatment response
Treatment failure | Through study completion, an average of 12 months
  TB Treatment failure during the study period.
TB recurrence | Through study completion, an average of 12 months
  TB recurrence during the study period
Number and severity of hepatic safety events | Through study completion, an average of 12 months
  Safety measures monitored throughout the study period.
Number and severity of adverse events (SAEs) | Through study completion, an average of 12 months
  Safety measures monitored throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wallis - Professor, Principal Investigator — Aurum Institute; Andrea Rachow, MD, Principal Investigator — LMU
Locations (1):
- MRC Unit The Gambia at LSHTM, Fajara, The Gambia, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available after the publication of the primary trial report. The end date has not yet been determined.
Access Criteria: Access will be available through the NIH TB Portals system.
URL: https://tbportals.niaid.nih.gov/

REFERENCES:
- [Background] Wallis RS, Sabi I, Lalashowi J, Bakuli A, Mapamba D, Olomi W, Siyame E, Ngaraguza B, Chimbe O, Charalambous S, Rachow A, Ivanova O, Zurba L, Myombe B, Kunambi R, Hoelscher M, Ntinginya N, Churchyard G. Adjunctive N-Acetylcysteine and Lung Function in Pulmonary Tuberculosis. NEJM Evid. 2024 Sep;3(9):EVIDoa2300332. doi: 10.1056/EVIDoa2300332. Epub 2024 Aug 27. PMID 39189858
- See also: TB Sequel website — https://www.tbsequel.org/